CLINICAL TRIAL: NCT02200094
Title: Micardis®. Observational Study
Brief Title: Micardis®. Observational Study in Patients With Essential Hypertension
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.361
Record Dates: First submitted 2014-07-24; First posted 2014-07-25 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Outpatients with essential hypertension
  Interventions: Drug: Low dose of Telmisartan, once daily; Drug: High dose of Telmisartan, once daily

INTERVENTIONS:
Drug: Low dose of Telmisartan, once daily
  Other Names: Micardis®
Drug: High dose of Telmisartan, once daily
  Other Names: Micardis®

SUMMARY:
This study is designed to supplement, under conditions of usual clinical practice, the data on the efficacy and safety of Micardis® collected during the clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex over the age of 18 years suffering from essential hypertension requiring treatment according to the physician

Exclusion Criteria:

* Hypersensitivity to the active component or to any of the excipients
* Pregnancy and lactation
* Biliary obstructive disorders
* Severe hepatic impairment
* Severe renal impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients over 18 years of age suffering essential hypertension, treated by general practitioners and/or specialists
Sampling Method: Non-Probability Sample
Enrollment: 4532 (Actual)
Dates: Start 1999-12; Primary Completion 2000-10 (Actual)

PRIMARY OUTCOMES:
Changes in systolic and diastolic blood pressure | Baseline, 4 weeks and 3 months after start of treatment
Percentage of patients with dose titration to 80 mg | 4 weeks and 3 months after start of treatment
Number of patients with adverse events | Up to 3 months after start of treatment
Global evaluation of treatment compliance by investigator, a 6-point rating scale | 4 weeks and 3 months after start of treatment